CLINICAL TRIAL: NCT05406427
Title: Monitorings the Physiological Mechanism of Airway Pressure Release Ventilation(APRV) in Acute Respiratory Distress Syndrome (ARDS) Patients by Electrical Impedance Tomography(EIT)
Brief Title: Monitorings the Physiological Mechanism of Airway Pressure Release Ventilation in ARDS Patients by EIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: EIT20220109
Record Dates: First submitted 2022-04-05; First posted 2022-06-06 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-06

CONDITIONS: Electrical Impedance Tomography; ARDS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Effects of airway pressure release ventilation on pulmonary ventilation, shunt and perfusion in patients with ARDS

DETAILED DESCRIPTION:
Effects of airway pressure release ventilation on respiratory mechanisms including ventilation distribution, intrapulmonary shunt and V/Q match in lungs of ARDS evaluated by EIT at different time points.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old < age < 80 years old
2. Diagnosed as moderate or severe ARDS according to the Berlin 2014 definition
3. Predicted APRV mechanical ventilation for more than 72 hours

Exclusion Criteria:

Excluded if any of the following exclusion criteria are met:

1. APRV contraindications such as pneumothorax, severe chronic obstructive pulmonary disease, severe asthma, intracranial hypertension
2. Pregnant women
3. Severe cardiac dysfunction (New York Heart Association class III or IV, acute coronary syndrome or sustained ventricular tachyarrhythmia), right heart enlargement due to chronic cardiopulmonary disease, cardiogenic shock or cardiac hand
4. Refractory shock
5. BMI>35

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Include as many subjects as possible according to the research protocol
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
tidal volume distribution during APRV at 24 hours after APRV | 24 hours after APRV mechanical ventilation
  we will use electrical impedance tomography(EIT) to monitor tidal volume distribution during APRV

SECONDARY OUTCOMES:
tidal volume distribution during APRV | Before APRV mechanical ventilation and 2, 6, 12, 48, 72 hours after APRV mechanical ventilation
  tidal volume distribution electrical impedance tomography(EIT) during APRV
Intrapulmonary shunt during APRV | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Intrapulmonary shunt percent represented regions that were only perfused calculated as the slope of regional impedance-time curves after saline bolus injection evaluated by EIT
V/Q match | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  V/Q match is monitored by EIT
tidal volume(Vt) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Vt is the volume of air inhaled or exhaled per breath during mechanical ventilation
Plateau pressure | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Plateau pressure is the airway pressure at the end of inspiratory pause
Positive end breath pressure | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Positive end breath pressure(PEEP) is the airway pressure at the end of each breath which is set by clinicians
Driving pressure(DP) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  DP=Plateau pressure-PEEP
Compliances(Cs) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Cs=DP/Vt
Peak pressure | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Peak pressure is the maximum pressure in the airway during ventilation occurs at the end of inspiration.
Mean pressure | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Mean pressure is the average airway pressure over a number of breathing cycles
Right ventricular area fractional change | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Right ventricular area fractional change is a simple and repeatable ultrasound method for evaluating right ventricular function. Methods: The right ventricular end-diastolic area (RVEDA) and right ventricular end- systolic area (RVESA) were measured on the apical four-chamber section by two-dimensional ultrasound. RVAC=(RVEDA- RVESA)/RVEDA*100%.
Tricuspid annular systolic displacement (TAPSE) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  TAPSE:Measurement method: TAPSE was measured on the four-chamber section of the apex of the heart by M-mode ultrasound. the sampling line was placed at the side wall of the tricuspid valve ring, parallel to the free wall of the right ventricle as far as possible, and the displacement of the tricuspid valve ring was measured from the end of diastole to the end of systole.
Tricuspid annular systolic S' velocity (TS') | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  TS' is an objective and accurate ultrasound technique for evaluating right ventricular function.Measurement method:The sample volume was applied to the free wall of the RV and the peak velocity of tricuspid annulus motion was measured in the four-chamber section of the apex by tissue doppler imaging (TDI).
Right ventricular end-diastolic area/left ventricular end-diastolic area (RVEDA/LVEDA) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  RVEDA/LVEDA a simple and repeatable ultrasound method for evaluating dynamics changes of right ventricular function.Methods: The right ventricular end-diastolic area (RVEDA) and left ventricular end-systolic area (LVEDA) were measured on the apical four-chamber section by two-dimensional ultrasound.
Pulmonary circulatory resistance (PVR) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  Increased PVR can lead to deterioration of RV function.Pulse Doppler imaging (PWD) was used to obtain the pulmonary artery flow spectrum from the pulmonic valve on the short axial section of the parasternal great vessels.
stroke volume index(SVI) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  SVI is monitored by two-dimension ultrasound
cardiac index (CI) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  The amount of blood pumped by the heart in liters per minute divided by the body surface area in square meters
Heart rate(HR) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  HR is one of the basic parameters of hemodynamics
Systolic blood pressure(SBP) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  SBP is one of the basic parameters of hemodynamics
Mean arterial pressure (MAP) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  MAP is one of the basic parameters of hemodynamics
Cardiac output(CO) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  The amount of blood expelled from one ventricle per minute
Stroke volume | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  The amount of blood expelled from one ventricle during a single cardiac beat
Arterial partial pressure of oxygen (PaO2) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  PaO2 is one of the key indicators of patients' respiratory status which can be obtained from arterial blood gas analysis.
Arterial partial pressure of carbon dioxide(PaCO2) | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  PaCO2 is one of the key indicators of pulmonary ventilation which can be obtained from arterial blood gas analysis.
oxygenation index | Before APRV mechanical ventilation and 2, 6, 12, 24, 48, 72 hours after APRV mechanical ventilation
  oxygenation index=PaO2/fraction of inspired oxygen
Sequential Organ Failure Assessment score | 2 hours within admission to ICU and 24 hours after inclusion in the study
  The higher the Sequential Organ Failure Assessment(SOFA) score(0~24), the higher the disease risk factor and the higher the mortality rate
Acute Physiology and Chronic Health Evaluation score | 2 hours within admission to ICU and 24 hours after inclusion in the study
  The higher the Acute Physiology and Chronic Health Evaluation(APACHE II) score(0~71), the higher the disease risk factor and the higher the mortality rate. In particular, the accuracy of group patient prediction is high.In particular, the accuracy of group patient prediction is high.
Duration of ventilation after randomization | from the day of randomization to the day of extubation or the day of death,assessed up to 90 days
  Time to mechanical ventilation in the ICU after randomization or time to mechanical ventilation after randomization until extubation or death
Mortality at 28 days after randomization | 28 days after the beginning of randomization
  Mortality at 28 days after randomization
ICU length of stay | the whole period of stay in ICU from the day of randomization to the day of discharge from ICU or the day of death,assessed up to 90 days
  Duration of ICU stay after randomization until surviving transfer out of ICU

CONTACTS AND LOCATIONS:
Overall Officials: xiaojing zou, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Y, Jin X, Lv Y, Wang P, Yang Y, Liang G, Wang B, Kang Y. Early application of airway pressure release ventilation may reduce the duration of mechanical ventilation in acute respiratory distress syndrome. Intensive Care Med. 2017 Nov;43(11):1648-1659. doi: 10.1007/s00134-017-4912-z. Epub 2017 Sep 22. PMID 28936695
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Mauri T, Spinelli E, Scotti E, Colussi G, Basile MC, Crotti S, Tubiolo D, Tagliabue P, Zanella A, Grasselli G, Pesenti A. Potential for Lung Recruitment and Ventilation-Perfusion Mismatch in Patients With the Acute Respiratory Distress Syndrome From Coronavirus Disease 2019. Crit Care Med. 2020 Aug;48(8):1129-1134. doi: 10.1097/CCM.0000000000004386. PMID 32697482
- [Result] Safaee Fakhr B, Araujo Morais CC, De Santis Santiago RR, Di Fenza R, Gibson LE, Restrepo PA, Chang MG, Bittner EA, Pinciroli R, Fintelmann FJ, Kacmarek RM, Berra L. Bedside monitoring of lung perfusion by electrical impedance tomography in the time of COVID-19. Br J Anaesth. 2020 Nov;125(5):e434-e436. doi: 10.1016/j.bja.2020.08.001. Epub 2020 Aug 7. No abstract available. PMID 32859359
- [Result] Kollisch-Singule M, Emr B, Smith B, Ruiz C, Roy S, Meng Q, Jain S, Satalin J, Snyder K, Ghosh A, Marx WH, Andrews P, Habashi N, Nieman GF, Gatto LA. Airway pressure release ventilation reduces conducting airway micro-strain in lung injury. J Am Coll Surg. 2014 Nov;219(5):968-76. doi: 10.1016/j.jamcollsurg.2014.09.011. Epub 2014 Sep 19. PMID 25440027

DOCUMENTS (1):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT05406427/Prot_000.pdf